CLINICAL TRIAL: NCT07166614
Title: Comparison of Respiratory and Hemodynamic Effects of Dexmedetomidine vs. Propofol in High-Risk Patients Undergoing ERCP: A Prospective Randomized Controlled Study
Brief Title: Dexmedetomidine vs Propofol in High-Risk ERCP Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hacer Sebnem Turk, associate professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: turk-25
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Depression; Hypoxemia; Hypotension Drug-Induced; Bradycardia
Keywords: Dexmedetomidine; propofol; adverse event; ERCP
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Hypotension; Bradycardia | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group d (Experimental): A loading dose of dexmedetomidine at 1 μg/kg was administered over 10 minutes prior to the procedure. During the procedure, an infusion at 0.5 μg/kg/h was maintained, which was discontinued at the end of the procedure
  Interventions: Drug: dexmedetomidin
- group p (Active Comparator): In our ERCP unit, induction was performed according to the standard protocol using fentanyl 1 µg/kg and propofol 1 mg/kg.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: dexmedetomidin — Dexmedetomidine is a highly selective α2-adrenergic receptor agonist with sedative, anxiolytic, and analgesic properties. Unlike many other sedatives, it provides sedation without significant respiratory depression, though it may cause bradycardia and hypotension
  Arms: group d
Drug: Propofol — Propofol is a short-acting intravenous anesthetic agent widely used for induction and maintenance of anesthesia as well as procedural sedation. It provides rapid onset and recovery, but is associated with respiratory depression and hypotension
  Arms: group p

SUMMARY:
ERCP requires deep sedation due to pain and discomfort, but propofol-commonly used with opioids-often causes respiratory and cardiovascular complications, especially in elderly or high-risk patients. Dexmedetomidine offers sedation without respiratory depression but may lower blood pressure and heart rate. Current monitoring often relies only on SpO₂, while capnography and the Integrated Pulmonary Index (IPI) provide earlier detection of respiratory events but are underused in ERCP studies.

This study compares dexmedetomidine and propofol in high-risk ERCP patients, focusing on respiratory and hemodynamic effects, propofol consumption, recovery, and discharge times. The hypothesis is that dexmedetomidine will cause fewer adverse respiratory and hemodynamic effects.

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is uncomfortable and painful for patients. Moreover, immobility is required for procedural success, which necessitates deep sedation. Recently, propofol combined with an opioid has been frequently used for this purpose . However, propofol is associated with respiratory depression, hypoxemia, and hypotension, leading to increased cardiopulmonary complications. These risks become more significant in elderly patients and those with high comorbidity. The use of alternative sedative agents or combinations aims to reduce propofol dosage and minimize cardiopulmonary complications.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist that reduces noradrenergic neuronal activity and is widely used for its sedative and anxiolytic properties. Unlike propofol, dexmedetomidine provides sedation without causing respiratory depression, even at loading doses. Several studies have evaluated the effects of dexmedetomidine and propofol on sedation in gastrointestinal endoscopic procedures . However, dexmedetomidine infusion alone has been shown to be less effective than propofol in terms of sedation quality, and it is associated with significant decreases in blood pressure and heart rate. These adverse events raise concerns regarding the use of dexmedetomidine in high-comorbidity patients requiring stable hemodynamics . Therefore, further studies are needed to evaluate the efficacy and safety of dexmedetomidine versus propofol in high-risk patients undergoing ERCP.

During endoscopy, monitoring of heart rate (HR), arterial blood pressure (BP), and pulse oximetry (SpO₂) is commonly used. Capnography with end-tidal CO₂ (ETCO₂) monitoring enables early detection of hypoventilation and apnea. Accordingly, both national and international guidelines (US and Europe) recommend capnography for monitoring during endoscopic procedures . The Integrated Pulmonary Index (IPI) incorporates HR, respiratory rate, SpO₂, and ETCO₂ parameters into an algorithm (14). It is considered the earliest method for detecting respiratory events and has been shown to be effective during endoscopic sedation.

However, studies evaluating the respiratory effects of sedative agents used in ERCP have been limited to SpO₂ values and adverse events, without assessment of ETCO₂ or IPI parameters.

In the study, the investigator primarily aimed to compare the respiratory and hemodynamic effects of dexmedetomidine versus propofol in high-risk patients undergoing ERCP. Secondarily, we evaluated total propofol consumption, recovery time, and discharge time from the endoscopy unit. Our hypothesis was that dexmedetomidine sedation in high-risk ERCP patients would result in fewer respiratory and hemodynamic side effects compared to propofol.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* ASA physical status III-IV
* scheduled for ERCP in the Gastroenterology Endoscopy Unit of our hospital

Exclusion Criteria:

* pregnant women;
* patients with neuropsychiatric disease,
* substance abuse, or known allergy to the sedatives used;
* patients with baseline heart rate ≤50 bpm;
* those who did not provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
heart rate | during the endoscopy (30-60 minute)
  heart rate
arterial blood pressure | during the endoscopy (30-60 minute)
  arterial blood pressure
oxygen saturation | during the endoscopy (30-60 minute)
  oxygen saturation
end-tidal CO₂ | during the endoscopy (30-60 minute)
  end-tidal CO₂

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli etfal research and training hospital, Sarıyer, Istanbul, Turkey (Türkiye)